CLINICAL TRIAL: NCT06174051
Title: The Effectiveness of Flashforward EMDR Treatment for Patients With an ICD
Brief Title: Flashforward EMDR Treatment for Patients With an ICD
Acronym: eFFective
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Leonieke Kranenburg, Associate professor, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 85546
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Anxiety and Fear
Keywords: EMDR; Flashforward; Anxiety; ICD
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: In this study, three groups are compared in a parallel setting. One group will receive EMDR following the flashforward procedure, one group will receive EMDR following the flashback procedure, and the last group will be on a wait list and fill out the questionnaires without receiving EMDR treatment.
Masking Description: The study will have an open label, since the care provider (the psychologist) needs to know which procedure to follow and the participants will understand in which group they are once the therapy start.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FF EMDR (Experimental): Subjects in this group will receive two EMDR treatment sessions following the flashforward protocol.
  Interventions: Behavioral: Flashforward EMDR
- FB EMDR (Active Comparator): Subjects in this group will receive two EMDR treatment sessions following the flashback protocol.
  Interventions: Behavioral: Flashback EMDR
- Control group (No Intervention): Subjects in this group will not receive any treatment until the wait list period (4 weeks) is over

INTERVENTIONS:
Behavioral: Flashforward EMDR — The Flashforward procedure in EMDR-treatment aims to reduce fear evoked by images of imagined future adverse events.
  Arms: FF EMDR
Behavioral: Flashback EMDR — The Flashback procedure in EMDR-treatment aims to successfuly process the memories of traumatic events that happened in the past.
  Arms: FB EMDR

SUMMARY:
The goal of this randomized controlled trial is to test whether flashforward (FF) EMDR alone is effective in reducing anxiety symptoms in patients with an implantable cardioverter defibrillator (ICD). Participants will fill out several questionnaires to asses their level of anxiety, depression symptoms and quality of life before, during and after treatment.

DETAILED DESCRIPTION:
Patients with an implantable cardioverter defibrillator (ICD) are at risk of ventricular arrhythmias (VA). The ICD is a device that can treat VA by antitachycardia pacing or ICD shocks. Since ICD shocks are painful and unpredictable, patients with an ICD can suffer from anxiety symptoms. Eye movement desensitization and reprocessing treatment (EMDR) is an effective treatment to enhance the process of traumatic events. In addition, this treatment has also shown to be able to reduce anxiety symptoms. EMDR treatment according to standard protocol starts with flashback (FB) procedure and may be followed by the flashforward (FF) procedure. The FB procedure focusses on events that happened in the past, while the FF procedure aims to reduce fear evoked by images of imagined future adverse events. So far, it is not clear whether the FB procedure is always necessary for the EMDR treatment to be effective. Moving straight towards application of the FF procedure (without first applying the FB procedure), may save treatment time and costs. Therefore, the main objective in this study is to test whether flashforward (FF) EMDR alone is effective in reducing anxiety symptoms in ICD patients. This will be tested with a pilot randomized controlled trial with a three-arm repeated measures design. Subjects will either receive FF EMDR, FB EMDR or no EMDR during the study. To measure their heart focussed anxiety, subjects will fill out the Cardiac Anxiety Questionnaire (CAQ) before, during and after treatment or waiting period.

ELIGIBILITY:
Inclusion Criteria:

* subjects have an ICD;
* subjects have clinical anxiety symptoms related to their ICD.

Exclusion Criteria:

* insufficient knowledge on Dutch or English language;
* severe psychiatric disorders that warrant (other) psychiatric first, such as suicidality or psychotic disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Cardiac Anxiety Questionnaire (CAQ) | Baseline (Before treatment T0), after the first treatment session T1(for wait list after 2 weeks), and after the second treatment session T2 (for wait list after 4 weeks)
  Self-report questionnaire to asses heart focussed anxiety

SECONDARY OUTCOMES:
PTSD Check-List (PCL-5) | Baseline (Before treatment T0) and after the second treatment session T2 (for wait list after 4 weeks)
  Self-report questionnaire to examine PTSD symptoms
General Anxiety Questionnaire (GAD-7) | Baseline (Before treatment T0) and after the second treatment session T2 (for wait list after 4 weeks)
  Self-report questionnaire to examine general anxiety symptoms
Patient Health Questionnaire (PHQ-9) | Baseline (Before treatment T0) and after the second treatment session T2 (for wait list after 4 weeks)
  Self-report questionnaire to examine depression symptoms
EuroQol (EQ5D-5L) | Baseline (Before treatment T0) and after the second treatment session T2 (for wait list after 4 weeks)
  Self-report questionnaire to examine quality of life

OTHER OUTCOMES:
Life Events Checklist (LEC-5) | Baseline (Before treatment T0)
  Self-report questionnaire to obtain information on previous traumatic life events

IPD SHARING:
Plan to Share IPD: No
Data will be available, anonymized, to other researchers, upon reasonable request.